CLINICAL TRIAL: NCT01720342
Title: Enable® Aortic Sutureless Bioprosthesis Evaluation: A Post-market Release Non-interventional Study
Brief Title: Enable® Aortic Sutureless Bioprosthesis Evaluation
Acronym: EASE
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Organization: Medtronic Cardiovascular (Industry)
Other Study IDs: EASE Enable
Record Dates: First submitted 2012-10-22; First posted 2012-11-02 (Estimated); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Aortic Valve Stenosis; Aortic Valve Insufficiency
Keywords: Medtronic Enable® aortic bioprosthesis; Aortic valve stenosis; Aortic valve insufficiency; "Real world" patients
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Aortic valve stenosis, aortic valve insufficiency: Patients with aortic valve insufficiency and/or aortic valve stenosis who require AVR.
  Interventions: Procedure: Aortic Valve Replacement surgery

INTERVENTIONS:
Procedure: Aortic Valve Replacement surgery — Aortic Valve Replacement surgery of the native aortic valve with the Enable® aortic bioprosthesis.
  Other Names: Medtronic ATS 3f Enable® Aortic Bioprosthesis (Model 6000)

SUMMARY:
The EASE Enable study is intended to collect additional data on the clinical outcomes of the Medtronic Enable® Aortic Bioprosthesis in "real world" patients.

DETAILED DESCRIPTION:
The EASE Enable study is intended to characterize the clinical performance of the Medtronic Enable® aortic bioprosthesis in a post-market real-world setting.

This is a Non-randomized, prospective, non-interventional multi-center post-market release (PMR) study. Up to 800 subjects will be enrolled at up to 40 centers in Europe. After aortic valve replacement with the Enable® aortic bioprosthesis, each patient will have routine follow-up visits at the following intervals: at 30 days post-implant (at 30 days post-implant or prior to hospital discharge, whatever comes first), within 6 months following implantation, 1 year and annually thereafter up to 5 years post-implant.

ELIGIBILITY:
Inclusion Criteria:

* Patient with aortic valve stenosis, aortic valve insufficiency or a combination of the two.
* Patient requires replacement of his/her native aortic valve with a bioprosthesis with or without concomitant procedures.
* Patient is above the minimum age as required by local regulations to be participating in a clinical study.
* Patient is willing to return to the implant site for follow-up visits.
* Patient has been adequately informed of this clinical study and is willing to sign the patient Data Release Form.

Exclusion Criteria:

* Patient requires replacement of two or more valves.
* Patient who underwent previous aortic valve replacement (AVR).
* Patient with native bicuspid aortic valve.
* Patient with active endocarditis or other systemic infection.
* Patient dilatation of the ascending aorta, deformations or irregular aortic annulus or ascending aorta geometry as seen via preoperative imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with aortic valve stenosis, aortic valve insufficiency or a combination of the two who require aortic valve replacement are eligible for this study, if they meet all study inclusion criteria and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2013-02; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Clinical performance during implant procedure, at 30 days post-implant (or prior to hospital discharge, whatever comes first), within 6 months post-operation, 1 year and annually thereafter up to 5 years post-procedure. | During implant procedure, at 30 days post-implant (or prior to hospital discharge, whatever comes first), within 6 months post-operation, 1 year and annually thereafter up to 5 years post-procedure.
  The early and late (up to five years) clinical performance of the Enable® aortic bioprosthesis will be characterized. Measures of clinical performance will include hemodynamic performance by echocardiography, New York Heart Association (NYHA) Functional Classification and safety (SAEs, ADEs, SADEs).

CONTACTS AND LOCATIONS:
Overall Officials: Otto Dapunt, MD, Principal Investigator — LKH Universitätsklinik Graz, Austria
Locations (17):
- France (2):
  - Centre Hospitalier Régional Universitaire de Lille (CHRU), Lille
  - Centre Hospitalier Universitaire de Saint-Etienne Hôpital Nord, Saint-Etienne
- Germany (6):
  - Universitätsklinikum Düsseldorf (UKD), Düsseldorf
  - Medizinische Hochschule Hannover (MHH), Hanover
  - Deutssches Herzzentrum Muenchen, Munich
  - Universitätsklinikum Münster (UKM), Münster
  - Klinikum Oldenburg GmbH, Oldenburg
  - Universitätsklinikum Ulm, Ulm
- Italy (3):
  - Casa Di Cura Privata 'Montevergine' S.p.A., Mercogliano
  - Ospedale Luigi Sacco, Milan
  - Azienda Complesso Ospedaliero S.Filippo Neri, Rome
- Netherlands (2):
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Leids Universitair Medisch Centrum, Leiden
- Spain (2):
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospiten Rambla, Santa Cruz de Tenerife
- Inselspital, Bern, Switzerland
- The James Cook University Hospital, Middlesbrough, United Kingdom

REFERENCES:
- [Background] Martens S, Sadowski J, Eckstein FS, Bartus K, Kapelak B, Sievers HH, Schlensak C, Carrel T. Clinical experience with the ATS 3f Enable(R) Sutureless Bioprosthesis. Eur J Cardiothorac Surg. 2011 Sep;40(3):749-55. doi: 10.1016/j.ejcts.2010.12.068. Epub 2011 Feb 20. PMID 21342776
- [Background] Englberger L, Carrel TP, Doss M, Sadowski J, Bartus K, Eckstein FF, Asch FM, Martens S. Clinical performance of a sutureless aortic bioprosthesis: five-year results of the 3f Enable long-term follow-up study. J Thorac Cardiovasc Surg. 2014 Oct;148(4):1681-7. doi: 10.1016/j.jtcvs.2014.03.054. Epub 2014 Apr 4. PMID 24787699